CLINICAL TRIAL: NCT02688452
Title: Water Oxygenation and Brain Activity: A Magnetoencephalographic (MEG) Pilot Study
Brief Title: Water Oxygenation and Brain Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 15-00230
Record Dates: First submitted 2016-02-03; First posted 2016-02-23 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Muscle Damage
Keywords: strenuous exercise; muscle soreness
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Young Healthy Adults
  Interventions: Dietary Supplement: Control Unmodified Placebo Water; Dietary Supplement: Electrokinetically modified water (EMW)
- Group 2 (Active Comparator): Young Healthy Adults
  Interventions: Dietary Supplement: Electrokinetically modified water (EMW); Dietary Supplement: Control Unmodified Placebo Water

INTERVENTIONS:
Dietary Supplement: Control Unmodified Placebo Water
  Arms: Group 1
Dietary Supplement: Electrokinetically modified water (EMW)
  Other Names: Reliant Recovery Water
  Arms: Group 1
Dietary Supplement: Electrokinetically modified water (EMW)
  Arms: Group 2
Dietary Supplement: Control Unmodified Placebo Water
  Arms: Group 2

SUMMARY:
The primary purpose of this interventional, placebo controlled, crossover, double blind, basic science exploratory study is to investigate whether there is a difference in brain electrophysiological oscillatory activity in healthy adults before and after oral consumption of water containing very small bubbles of oxygen (electrokinetically modified water).

ELIGIBILITY:
Inclusion Criteria:

* Men or women of any ethnic background;
* living in New York tri-state area;
* fluent in English;
* normal or corrected to normal vision and hearing;
* willing to complete all study procedures; and
* capable of giving written informed consent.

Exclusion Criteria:

* A history of gross brain abnormalities such as stroke, severe ventriculomegaly or severe periventricular white matter abnormalities;
* a history of serious psychiatric or neurological disorders, including psychosis or major depression, alcohol or drug abuse, brain injury, seizure disorder, brain tumor, etc.;
* taking psychoactive medications, including antipsychotics, anxiolytics and antidepressants, or cognitive enhancers such as cholinesterase inhibitors;
* presence of contraindications for MEG or MRI recording, including any of the following: cardiac pacemaker, intracranial clips, metal implants, or external clips within 10 mm of the head, metal in eyes, claustrophobia, obesity and/or any other reason leading to difficulty staying in the MEG or MRI for up to one hour.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in spectral properties measured before and after drinking the test products using Magnetoencephalography (MEG) measurements | 1 Week
  Magnetic fields will be recorded using a 275-channel whole-head MEG system
Changes in localization of spontaneous brain activity measured before and after drinking the test products using Magnetoencephalography (MEG) measurements | 1 Week
  Magnetic fields will be recorded using a 275-channel whole-head MEG system

SECONDARY OUTCOMES:
Self reported changes in behavioral state before and after drinking test product | 1 Week

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Llinás, MD, PhD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States